CLINICAL TRIAL: NCT01822119
Title: Clinical Performance of a Transcutaneous Bone Conduction Hearing Solution (Baha® Attract System). A Multicentre, Open, Prospective Clinical Investigation. 3 Months Investigation With a 6 Months Follow-up
Brief Title: Clinical Performance of a Transcutaneous Bone Conduction Hearing Solution (Baha® Attract System)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5484
Record Dates: First submitted 2013-03-19; First posted 2013-04-02 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Deafness; Hearing Loss; Hearing Loss, Conductive
MeSH Terms: conditions — Deafness; Hearing Loss; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baha Attract System (Experimental): This transcutaneous solution is based on a magnet coupling using magnets on both side of the skin;
  * One implant magnet
  * One external magnet on which a sound processor is attached, i.e. the Sound Processor magnet (SP magnet)
  Interventions: Device: Baha Attract System

INTERVENTIONS:
Device: Baha Attract System

SUMMARY:
The rationale behind this clinical performance investigation is to collect data regarding the usability of the Baha Attract System in patients with hearing impairment that are candidates for Baha surgery:

* To describe the expected hearing performance with the Baha Attract in comparison to unaided hearing thresholds or a pre-test situation using a sound processor together with a softband
* Which sound processor to select, i.e. BP100 vs BP110
* Improve the fitting process for the sound processor
* Selection of sound processor magnet at time of fitting and over time

ELIGIBILITY:
Inclusion Criteria:

* Conductive hearing loss in the implanted ear. Bone conduction thresholds with a pure tone average of 500, 1000, 2000 and 3000 Hz <30 decibel (dB) hearing level (HL)
* Single-sided Sensorineural Deafness (SSD). Bone conduction thresholds with a pure tone average of 500, 1000, 2000 and 3000 Hz <30 dB hearing level (HL) in the best ear
* Signed informed consent

Exclusion Criteria:

* Uncontrolled diabetes as judged by the investigator
* Condition that could jeopardize osseointegration and/or wound healing, e.g. osteoporosis, psoriasis and use of corticosteroids
* Unable to follow investigational procedures, e.g. to complete quality of life scales
* Less than 4mm of soft tissue pre-operatively
* Participation in another investigation with pharmaceuticals and/or device
* Condition that may have an impact on the outcome of the investigation as judged by the investigator
* Subjects that have received radiation therapy at the same side of the skull where the Baha Attract will be positioned
* Suitable implant position for the Baha BI300 implant system (4 mm and 3 mm) not found during surgery due to insufficient bone quality and/or bone thickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, A/Professor, Principal Investigator — The HEARing CRC & HearWorks, University of Melbourne
Locations (4):
- The HEARing CRC & HearWorks, University of Melbourne, Melbourne, Victoria, Australia
- Clinica Las Condes, Santiago, Chile
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Bnai Zion MedicalCenter, Haifa, Israel

REFERENCES:
- [Result] Briggs R, Van Hasselt A, Luntz M, Goycoolea M, Wigren S, Weber P, Smeds H, Flynn M, Cowan R. Clinical performance of a new magnetic bone conduction hearing implant system: results from a prospective, multicenter, clinical investigation. Otol Neurotol. 2015 Jun;36(5):834-41. doi: 10.1097/MAO.0000000000000712. PMID 25634465

RESULTS

PARTICIPANT FLOW:
Groups:
- Baha Attract System: This transcutaneous solution is based on a magnet coupling using magnets on both side of the skin;
  * One implant magnet
  * One external magnet on which a sound processor is attached, i.e. the Sound Processor magnet (SP magnet)
  Baha Attract System
Period: Overall Study
Arm/Group | Baha Attract System
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.8)
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Region of Enrollment [Number; unit: participants]
  Hong Kong | 8
  Israel | 6
  Australia | 8
  Chile | 5
Type of hearing loss [Number; unit: participants]
  Conductive hearing loss | 17
  Single-sided sensorineural deafness | 10

OUTCOME MEASURES:

1. Primary Outcome: Hearing Performance, PTA4 at 12 Weeks
Description: The change in pure-tone thresholds in free field measured by the difference in pure tone average PTA4 (Mean of thresholds at 500, 1000, 2000 and 4000 Hz) from the pre-operative unaided condition to the aided situation with the Baha Attract System at week 12.
Time Frame: Baseline before surgery and 12 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB | -18.4 (6.7)
Statistical Analysis 1: Comparison: Baha Attract System; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation

2. Primary Outcome: Hearing Performance, PTA4 at 36 Weeks
Description: The change in pure-tone thresholds in free field measured by the difference in pure tone average PTA4 (Mean of thresholds at 500, 1000, 2000 and 4000 Hz) from the pre-operative unaided condition to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB | -18.4 (6.9)
Statistical Analysis 1: Comparison: Baha Attract System; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation

3. Secondary Outcome: Hearing Performance, Individual Frequencies
Description: The change in pure-tone thresholds in free field measured by the difference at individual frequencies from the pre-operative unaided condition to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB
  Change in hearing level at 500HZ | -20.2 (14.4)
  Change in hearing level at 1000HZ | -25.2 (8.4)
  Change in hearing level at 2000HZ | -18.3 (9.5)
  Change in hearing level at 3000HZ | -18.7 (14.7)
  Change in hearing level at 4000HZ | -9.8 (10.8)
  Change in hearing level at 6000HZ | -5.0 (12.3)
  Change in hearing level at 8000HZ | -4.2 (10.7)
Statistical Analysis 1: Comparison: Baha Attract System; Statistically significant changes with the same value at 500 to 4000Hz; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; Change at 6000Hz; Test type: Superiority or Other; p = 0.0499, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; Change at 8000Hz; Test type: Superiority or Other; p = 0.0632, Fisher's non-parametric permutation test

4. Secondary Outcome: Hearing Performance, PTA4, Sound Processor on Softband Versus Baha Attract at 36 Weeks
Description: The change in pure-tone thresholds in free field measured by the difference in pure tone average PTA4 (Mean of thresholds at 500, 1000, 2000 and 4000 Hz) from the pre-operative aided situation with the Sound Processor on a softband to the aided situation with Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB | 0.926 (5.553)
Statistical Analysis 1: Comparison: Baha Attract System; Test type: Superiority or Other; p = 0.39, Fisher's non-parametric permutation test

5. Secondary Outcome: Hearing Performance, Individual Frequencies, Sound Processor on Softband Versus Baha Attract at 36 Weeks
Description: The change in pure-tone thresholds in free field measured by the difference in hearing levels of individual frequencies from the pre-operative aided situation with the Sound Processor on a softband to the aided situation with Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB
  500Hz | -0.741 (13.637)
  1000Hz | -1.67 (7.34)
  2000Hz | 1.67 (7.07)
  3000Hz | -0.37 (8.077)
  4000Hz | 4.44 (9.64)
  6000Hz | 6.92 (12.34)
  8000 | 3.80 (12.10)
Statistical Analysis 1: Comparison: Baha Attract System; 500Hz; Test type: Superiority or Other; p = 0.79, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 1000Hz; Test type: Superiority or Other; p = 0.26, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 2000Hz; Test type: Superiority or Other; p = 0.24, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 3000Hz; Test type: Superiority or Other; p = 0.83, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 4000Hz; Test type: Superiority or Other; p = 0.026, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 6000Hz; Test type: Superiority or Other; p = 0.0085, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 8000Hz; Test type: Superiority or Other; p = 0.13, Fisher's non-parametric permutation test

6. Secondary Outcome: Hearing Performance, Speech in Quiet, Unaided Versus Baha Attract at 36 Weeks
Description: The change in hearing performance, speech in quiet from the pre-operative unaided condition to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: % perception of presented words
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
% perception of presented words
  Change at 50dB presentation level | 50 (23.7)
  Change at 65dB presentation level | 46.4 (31.7)
  Change at 80dB presentation level | 24.2 (25.6)
Statistical Analysis 1: Comparison: Baha Attract System; Statistically significant improvement with the same value at all presentation levels; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

7. Secondary Outcome: Hearing Performance, Speech in Quiet, Aided With the Sound Processor on a Softband Versus Baha Attract at 36 Weeks
Description: The change in hearing performance, speech in quiet from the pre-operative aided situation with the Sond Processor on a softband to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: % perception of presented words
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
% perception of presented words
  Change at 50dB presentation level | 2.83 (23.80)
  Change at 65dB presentation level | 0.98 (13.49)
  Change at 80dB presentation level | 1.71 (7.80)
Statistical Analysis 1: Comparison: Baha Attract System; 50dB; Test type: Superiority or Other; p = 0.55, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 60dB; Test type: Superiority or Other; p = 0.72, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 80dB; Test type: Superiority or Other; p = 0.28, Fisher's non-parametric permutation test

8. Secondary Outcome: Hearing Performance, Speech in Noise, Unaided Versus Baha Attract at 36 Weeks
Description: The change in hearing performance, speech in noise from the pre-operative unaided condition to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: Signal to noise ratio
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
Signal to noise ratio | -15.0 (12.8)
Statistical Analysis 1: Comparison: Baha Attract System; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

9. Secondary Outcome: Hearing Performance, Speech in Noise, Aided With the Sound Processor on a Softband Versus Baha Attract at 36 Weeks
Description: The change in hearing performance, speech in noise from the pre-operative aided situation with the Sond Processor on a softband to the aided situation with the Baha Attract System at week 36.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: Signal to noise ratio
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
Signal to noise ratio | -3.79 (6.96)
Statistical Analysis 1: Comparison: Baha Attract System; Test type: Superiority or Other; p = 0.0092, Fisher's non-parametric permutation test

10. Secondary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: Change of APHAB scoring from the unaided pre-operative situation to the aided situation with Baha Attract at 36 weeks. APHAB questionnaire is a 24-item self-assessment inventory that evaluates the benefit experienced by the patient when using hearing amplification compared to the unaided situation. APHAB produces a Global score and scores for four subscales: ease of communication (EC), reverberation (RV), background noise (BN), and aversiveness (AV). The absolute APHAB scale is between 0 and 100%, where 0% indicates no problem and 100% indicates always problem. The change from unaided to aided hearing is presented. A positive value indicates an improvement, a negative value an impairment. This scale applies to all reported scores.
Time Frame: Baseline before surgery and 36 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
units on a scale
  Aversiveness | -4.04 (36.03)
  Ease of communication | 4.23 (52.16)
  Reverberation | 5.10 (42.78)
  Background noise | 8.92 (48.07)
  Global score | 6.76 (45.92)
Statistical Analysis 1: Comparison: Baha Attract System; Aversiveness; Test type: Superiority or Other; p = 0.59, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; Ease of Communication; Test type: Superiority or Other; p = 0.71, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; Reverberation; Test type: Superiority or Other; p = 0.59, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; Background noise; Test type: Superiority or Other; p = 0.40, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; Global score; Test type: Superiority or Other; p = 0.50, Fisher's non-parametric permutation test

11. Other Pre Specified Outcome: Time to Perform Surgery
Time Frame: Visit 2 (surgery)
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
minutes | 45.0 (14.6)

12. Other Pre Specified Outcome: Tissue Reduction Performed During Surgery
Description: Surgical thinning of the soft tissue flap was advocated when the soft tissue thickness exceeded 6 mm.
Time Frame: Visit 2 (surgery)
Population: Intention-to-Treat population, includes all patients who received surgical intervention.
Measure: Number; unit: participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
participants
  No tissue reduction | 24
  Tissue reduction | 3

13. Other Pre Specified Outcome: Implant Stability
Description: Implant Stability Quotient - ISQ, a scale from 1 to 100, where 100 represent the highest stability.
Time Frame: Visit 2 (surgery)
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
units on a scale | 75.7 (8.8)

14. Other Pre Specified Outcome: Choice of Sound Processor
Description: Type of sound processors BP100 and BP110 attached to a soft band (subject preference)
Time Frame: Baseline
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Number; unit: participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
participants
  BP100 | 6
  BP110 | 21

15. Other Pre Specified Outcome: Feedback Measurement, BP100
Description: Difference between softband measurement at visit 1 and measurement with the Baha Attract system at visit 6. Feedback is a measure of how much sound from the actuator (vibrator) returns to the microphones thus creating a loop of sound which sounds like high pitch noise. Measuring this is a part of the performance of the system, i.e how much gain can the sound processor produce before feedback occurs. Unit of measure is dB re output. A negative value of the change means less feedback.
Time Frame: Baseline before surgery and 12 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB
  400Hz | -13.2 (7.8)
  500Hz | -6.54 (3.98)
  630Hz | -4.29 (8.56)
  800Hz | -7.11 (6.84)
  1000Hz | -7.85 (4.59)
  1250Hz | -10.1 (2.4)
  1600Hz | -7.44 (2.88)
  2000Hz | -2.82 (1.59)
  2500Hz | -2.91 (3.64)
  3150Hz | -1.21 (3.66)
  4000Hz | 1.83 (3.42)
  5000Hz | 0.17 (4.37)
  6300Hz | 7.28 (7.62)
  8000Hz | 3.95 (3.26)

16. Other Pre Specified Outcome: Feedback Measurement, BP110
Description: as for outcome 15
Time Frame: Baseline before surgery and 12 weeks after surgery
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
dB
  400Hz | -3.50 (8.36)
  500Hz | -3.86 (8.46)
  630Hz | -4.20 (10.59)
  800Hz | -3.39 (9.16)
  1000Hz | -5.03 (7.17)
  1250Hz | -8.10 (7.87)
  1600Hz | -8.85 (6.51)
  2000Hz | -4.73 (4.65)
  2500Hz | -3.08 (4.10)
  3150Hz | -3.00 (3.30)
  4000Hz | 0.69 (4.86)
  5000Hz | 6.58 (6.24)
  6300Hz | 10.3 (4.7)
  8000Hz | 12.2 (9.7)

17. Other Pre Specified Outcome: Magnetic Force
Description: To investigate if the magnetic force required for sound processor magnet retention will change over time
Time Frame: Week 4, 6, 12 and 36
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
Newton
  4 weeks | 0.97 (0.30)
  6 weeks | 1.05 (0.37)
  12 weeks | 0.98 (0.29)
  36 weeks | 0.97 (0.28)

18. Other Pre Specified Outcome: Safety; Skin Evaluation
Description: Evaluation of the skin using the Patient and Observer Scar Assessment Scale (POSASa scale from 1 (normal skin) to 10 (worst scar imaginable).
Time Frame: 36 weeks
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
units on a scale
  Overall opinion observer | 1.52 (0.93)
  Overall opinion patient | 1.81 (1.21)

19. Other Pre Specified Outcome: Safety; Pain
Description: Evaluation of neuropathic pain or pain in the scar the last week by asking the patients to rate their experience on a scale from 1 (no, not at all) to 10 (yes, very much).
Time Frame: 36 weeks
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
units on a scale
  Neuropathic pain | 1.19 (0.79)
  Pain in the scar | 1.15 (0.77)

20. Other Pre Specified Outcome: Safety; Numbness
Description: Evaluation of numbness by asking the patients if they had experienced any numbness within 2 cm from the centre of the implant magnet or within and beyond 2 cm from the centre of the implant magnet.
Time Frame: 36 weeks
Population: Intention-to-Treat (ITT) population, includes all patients who received surgical intervention.
Measure: Number; unit: participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 27
participants
  No numbness | 21
  Numbness within 2 cm | 1
  Numbness within 2 cm and beyond | 5

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Baha Attract System
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 8/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baha Attract System (N=27)
Postoperative wound infection (Infections and infestations) | 2 (2)
Post procedural heamatoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baha Attract System (N=27)
Application site pain (General disorders) | 4 (4)
Implant site erythema (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days